CLINICAL TRIAL: NCT05042544
Title: The National Australian HCV Point-of-Care Testing Program: An Observational Cohort Study to Evaluate the Use of Finger-stick Point-of-care Hepatitis C Testing to Enhance Diagnosis and Treatment of HCV Infection
Brief Title: The National Australian HCV Point-of-Care Testing Program
Status: Recruiting | Type: Observational
Sponsor: Kirby Institute (Other Government)
Collaborators: Flinders University (Other)
Responsible Party: Sponsor
Other Study IDs: VHCRP2101
Record Dates: First submitted 2021-08-20; First posted 2021-09-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Hepatitis C
Keywords: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People at risk of HCV acquisition: This is an observational cohort study. Participants will be recruited from settings that provide services to people with a risk factor for the acquisition of HCV infection. Participants will attend a single visit to receive point-of-care HCV testing and complete a self-administered survey. Testing will be performed using point-of-care HCV antibody testing (results within 1-20 minutes, depending on the test) and if positive, HCV RNA testing will be performed. Participants who have previously had HCV infection or previously received HCV treatment will be tested using point-of-care HCV RNA testing. Participants will not receive treatment as a part of this study. Participants who are HCV RNA detectable will be linked to standard of care for any other clinical assessments and treatment initiation.
  Interventions: Diagnostic Test: Point-of-Care Testing

INTERVENTIONS:
Diagnostic Test: Point-of-Care Testing — Participants will be offered finger-stick point-of-care testing for HCV

SUMMARY:
The National Australian HCV Point-of-Care Testing Program will establish an observational cohort to evaluate whether scale-up of finger-stick point-of-care HCV testing increases diagnosis and treatment for HCV infection. Participants will be recruited from settings providing services to people with a risk factor for the acquisition of HCV infection (including drug treatment clinics, needle and syringe programs, homelessness settings, mental health services, prisons, and mobile outreach). Participants will attend a single visit to have their HCV RNA status tested and complete a self-administered survey. Participants will not receive treatment as a part of this study. Participants who are HCV RNA positive will be linked to standard of care.

DETAILED DESCRIPTION:
The advent of simple direct-acting antiviral hepatitis C (HCV) therapies with cure rates >95% is one of the greatest medical advances in decades, having led to a reversal in liver-related mortality. In Australia, treatment uptake has declined between 2016 (32,000 treated) and 2019/20 (2019: 11,500; 2020: 8,500).1 Progress towards HCV elimination has been impeded by COVID-19, affecting the delivery of national and state-based HCV strategies. Improving HCV treatment uptake to reduce disease burden is a key aim of global, national and state-based HCV strategies.2-4

Scale-up of HCV testing and treatment will be required to achieve elimination by 2030. Current diagnostic pathways require multiple visits to a practitioner reducing the proportion who receive a diagnosis. In Australia, 81% of people have had HCV antibody testing (indicates exposure), but only 47% have been HCV RNA tested (indicates active infection and the need for HCV treatment).5 Mathematical modelling suggests that HCV RNA testing needs to increase by at least 50% annually to achieve elimination in Australia by 2030.6

The Kirby Institute is an international leader in research evaluating the Xpert HCV assay (Grebely Lancet Gastro Hep 2017), having built a large network of Xpert platforms for HCV testing in needle and syringe programs, prisons, drug treatment clinics, tertiary hospitals, and Aboriginal Community Controlled Health Service. In Kirby-led research, point-of-care HCV testing interventions in needle and syringe programs and prisons have resulted in high HCV treatment uptake (70-90%). The Kirby Institute and Flinders University also have a strong track record of implementing point-of-care testing for STIs and COVID-19, providing an ideal foundation to scale-up Xpert HCV testing in Australia.

The Kirby Institute and Flinders University will establish the Australian National HCV Point-of-care Testing Program for the scale-up of point-of-care HCV RNA testing in services with high prevalence of HCV infection, including community health centres, drug treatment clinics, needle and syringe programs, and prisons. This program will include the development of standard operating procedures, logistics/deployment, initial set-up, an operator training program, and quality assurance and competency assessment program.

An observational cohort study that will be established to evaluate HCV treatment uptake following scale-up of point-of-care HCV testing among people with a risk factor for acquisition of HCV infection or people attending a service caring for people with risk factors for the acquisition of HCV infection. This study will also include the linkage of survey data to a range of administrative datasets which will be used to evaluate the impact of HCV testing and treatment scale-up on a range of long-term health outcomes.

Participants will be recruited from settings that provide services to people with a risk factor for the acquisition of HCV infection. Participants will attend a single visit to receive point-of-care HCV testing and complete a self-administered survey. Testing will be performed using point-of-care HCV antibody testing (results within 1-20 minutes, depending on the test) and if positive, HCV RNA testing will be performed. Participants who have previously had HCV infection or previously received HCV treatment will be tested using point-of-care HCV RNA testing. Participants will not receive treatment as a part of this study. Participants who are HCV RNA detectable will be linked to standard of care for any other clinical assessments and treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

1. Provided informed consent.
2. ≥ 18 years of age.
3. Have a risk factor for the acquisition of HCV infection (including current or past injecting drug use, previous incarceration, HIV infection, receiving blood products prior to 1990, having a tattoo or piercing in an unregulated environment, a needle-stick injury, or a mother with HCV).

   OR:
4. Are attending a service caring for people with risk factors for the acquisition of HCV infection (e.g. drug treatment clinics, needle and syringe programs, prisons, mobile outreach services, community health services, mental health services, and homelessness services).

Exclusion Criteria:

a. Is unable or unwilling to provide informed consent or abide by the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from settings that provide services to people with a risk factor for the acquisition of HCV infection, including drug treatment clinics, needle and syringe programs, prisons, mobile outreach services, community health services, mental health services, homelessness services, and other appropriate settings nationally. It is anticipated approximately 40,000 participants will be screened for HCV infection using point-of-care HCV testing.
Sampling Method: Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the proportion of HCV infected (HCV RNA quantifiable) participants who initiate HCV treatment at 12 weeks following HCV RNA testing. | 12 Weeks from enrolment
  HCV treatment

SECONDARY OUTCOMES:
To evaluate the proportion of people who accept point-of-care testing among those offered testing. | Recruitment phase
  Accepting testing
To evaluate the prevalence of current HCV infection (HCV RNA quantifiable) among people tested. | Recruitment phase
  Prevalence
To evaluate the time to HCV treatment uptake among HCV RNA detectable participants following HCV RNA testing | 52 weeks
  Time to treatment
To evaluate the proportion of HCV RNA detectable participants who initiate HCV treatment at 12 months (52 weeks) following detectable finger-stick point-of-care HCV RNA testing. | 52 weeks
  Initiation of treatment
To evaluate the proportion of participants who complete HCV direct-acting antiviral (DAA) treatment. | 52 weeks
  Completion of treatment
To evaluate the proportion of participants who achieve an SVR (defined as HCV RNA below the lower limit of quantitation at post treatment week 12) following a detectable HCV RNA test result. | 12 weeks
  SVR
To evaluate the proportion of participants who are HCV RNA negative at 12 months (52 weeks) following a detectable HCV RNA test. | 52 weeks
  HCV negative
To evaluate the cost-effectiveness of different testing strategies | 52 weeks
  Cost-effectiveness

CONTACTS AND LOCATIONS:
Locations (56):
- Australia (56):
  - Hepatitis ACT, Canberra, Australian Capital Territory
  - Western NSW LHD, Bathurst, New South Wales
  - Far West LHD, Broken Hill, New South Wales
  - Maari Ma Health Aboriginal Corporation, Broken Hill, New South Wales
  - Galambila Aboriginal Health Service, Coffs Harbour, New South Wales
  - Central Coast LHD, Gosford, New South Wales
  - Armajun Health Service Aboriginal Corporation, Inverell, New South Wales
  - Rekindling the Spirit Health Service, Lismore, New South Wales
  - Nepean Blue Mountains LHD, Penrith, New South Wales
  - North and Mid North Coast LHD, Port Macquarie, New South Wales
  - Walhallow Aboriginal Corporation, Quirindi, New South Wales
  - Bulgarr Ngaru Medical Aboriginal Corporation, South Grafton, New South Wales
  - Kirketon Road Centre, Sydney, New South Wales
  - NSLHD, Sydney, New South Wales
  - WSLHD Drug Health, Sydney, New South Wales
  - South West Sydney LHD, Sydney, New South Wales
  - Hepatitis NSW, Sydney, New South Wales
  - NSW Users and AIDS Association, Sydney, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - SESLHD Community and Mental Health POCT Allicance (SCAMPA), Sydney, New South Wales
  - SESLHD Drug Health, Sydney, New South Wales
  - Storr Liver Clinic (Westmead Hospital), Sydney, New South Wales
  - Sydney Local Health District, Sydney, New South Wales
  - Murrumbidgee & Southern LHD, Wagga Wagga, New South Wales
  - Hunter New England LHD, Waratah, New South Wales
  - ISLHD Drug and Alcohol Service, Wollongong, New South Wales
  - ADSCA - Alice Springs Hospital, Alice Springs, Northern Territory
  - Alcohol and Harm Reduction Biala, Brisbane, Queensland
  - Micah Projects, Brisbane, Queensland
  - Cairns Sexual Health Service, Cairns, Queensland
  - Hepatitis QLD, Coorparoo, Queensland
  - Kombi Clinic, Inala, Queensland
  - Metro South Addiction Services - Inala ADS, Inala, Queensland
  - Ipswich AODS, Ipswich, Queensland
  - Ipswich Sexual Health and BBV Service, West Moreton Health, Ipswich, Queensland
  - OneBridge, Maroochydore, Queensland
  - Central Adelaide Local Health Network, Adelaide, South Australia
  - Drug and Alcohol Services South Australia, Adelaide, South Australia
  - North Adelaide Local Health Network, Adelaide, South Australia
  - South Adelaide Local Health Network, Adelaide, South Australia
  - Hepatitis SA, Hackney, South Australia
  - Pangula Mannamurna Aboriginal Corporation, Mount Gambier, South Australia
  - Clinic 60 (Sexual Health Services), Hobart, Tasmania
  - Moreton Group Rural Health, New Town, Tasmania
  - Western Health, Footscray, Victoria
  - Eastern Health, Melbourne, Victoria
  - St Vincent's Hospital (Melbourne), Melbourne, Victoria
  - Youth Projects - The Living Room, Melbourne, Victoria
  - Latrobe Community Health Service Liited, Morwell, Victoria
  - Peer Based Harm Reduction Bunbury, Bunbury, Western Australia
  - South Terrace Clinic - Fremantle Hospital, Fremantle, Western Australia
  - Peer Based Harm Reduction WA, Perth, Western Australia
  - Hepatitis WA, Perth, Western Australia
  - Next Step East Perth, Perth, Western Australia
  - Next Step Fremantle, Perth, Western Australia
  - Next Step Warwick, Perth, Western Australia